CLINICAL TRIAL: NCT06493292
Title: Comparison of the Efficacy of Drug-Coated Balloons and Cutting Balloons in the Treatment of Autologous Arteriovenous Fistula Stenosis: A Multi-Center Prospective Real-World Study.
Brief Title: Effectiveness of Endoluminal Treatment of Autologous Arteriovenous Endovascular Fistula Failure
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Drug-Coated/Cutting Balloons
Record Dates: First submitted 2024-07-02; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Hemodialysis Access Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Endovascular therapy — Endovascular therapy is a minimally invasive interventional approach that utilizes the vascular system as a pathway to access and treat various pathological conditions within the body. By employing specialized catheters and devices, endovascular techniques enable precise delivery of therapeutic agents or interventional procedures directly to the target site, without the need for conventional open surgery.

SUMMARY:
This study was aimed at comparing the efficacy and safety of cutting balloons versus drug-coated balloons in treating venous segment stenosis of autologous arteriovenous fistulas.This is a prospective, multi-center cohort study.

DETAILED DESCRIPTION:
The study will recruit 180 patients with venous segment stenosis of autologous arteriovenous fistulas at multiple centers from June 2024 to December 2025. Patients will be divided into two cohorts based on the treatment method: the Cutting Balloon group and the Drug-Coated Balloon group. The primary outcomes observed will be the primary patency rates of the target lesion at 1, 3, 6, and 12 months post-operation, re-intervention rates of the target vessel, and the technical success rates and procedural success rates of the two devices, along with major adverse events during the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18 and 75 years.
2. Subjects possess a mature upper limb autologous arteriovenous fistula (AVF) and have undergone at least one hemodialysis session.
3. Target lesion must be located in the venous segment of the upper limb AVF.
4. Doppler ultrasound confirms that the target lesion stenosis is ≥50%, accompanied by at least one of the following clinical manifestations: elevated venous pressure during dialysis, abnormal fistula signs, significant reduction in blood flow (<200ml/min).
5. Guidewire and balloon successfully pass through the lesion and complete dilation. 6.Subjects or their legal representatives must understand the purpose of the trial, voluntarily participate in the clinical trial, and sign an informed consent form, while also being willing to adhere to the specific follow-up schedules set by this trial.

Exclusion Criteria:

1. Target lesion located in the arterial segment or anastomosis of the AVF.
2. Target lesion located in the lower limb AVF.
3. Subjects with previous stent implantation in the AVF.
4. Patients diagnosed with symptomatic central venous occlusive disease: AVF flow reduction accompanied by swelling of the ipsilateral limb, chest, or facial area, with DSA confirmation of central venous occlusive disease.
5. Subjects with two or more target lesions in the AVF (when two stenoses are less than 3 cm apart, they are considered as one target lesion).
6. Subjects with acute thrombosis in the AVF or who have undergone AVF thrombolysis or thrombectomy within the past 30 days.
7. Subjects who have undergone or plan to undergo surgical intervention on the AVF within 30 days.
8. Subjects with AVF infection or concurrent systemic active infection.
9. Subjects planning renal transplantation or switching to peritoneal dialysis within the next 12 months.
10. Subjects with diseases causing coagulopathy, such as thrombocytopenic purpura.
11. Subjects undergoing immunotherapy or suspected/diagnosed with vasculitis.
12. Subjects with allergies or contraindications to heparin or contrast agents.
13. Subjects who are pregnant or breastfeeding.
14. Subjects with a life expectancy of less than 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dysfunctional autogenous arteriovenous fistula patient: A stenosis in a hemodialysis access with significant hemodynamic changes: Based on angiography/ultrasound evaluation, the target lesion stenosis is ≥50%, and is accompanied by one or more of the following clinical and physiological abnormalities: natural fistula blood flow <480ml/min; unable to meet the required blood flow for the dialysis prescription; thrombosis in the autogenous arteriovenous fistula; elevated venous pressure during dialysis; difficult cannulation; decreased dialysis adequacy; and abnormal signs in the fistula, etc.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinically-driven target lesion re-intervention | 1-month#3-month#6-month#12-month
  Clinically-driven target lesion re-intervention refers to a repeat procedure performed on a previously treated lesion due to the recurrence of symptoms or other clinical indications, rather than being routinely scheduled.

SECONDARY OUTCOMES:
Target lesion primary patency | 1-month#3-month#6-month#12-month
  Target lesion primary patency refers to the treated lesion site remaining open and unobstructed without the need for any additional revascularization procedure during the follow-up period.
Target lesion assisted primary patency | 1-month#3-month#6-month#12-month
  Target lesion assisted primary patency refers to the treated lesion site remaining patent (open) during the follow-up period, but requiring an additional revascularization procedure, such as percutaneous transluminal angioplasty, to maintain patency of the target lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ye, Study Director — The Second Hospital of Nanjing Medical University; Pei Wang, Study Director — The First Affiliated Hospital of Zhengzhou University; Lan Zhang, Principal Investigator — Shanghai Jiao Tong University School of Medicine，Renji Hospital
Locations (3):
- China (3):
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Renji Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided